CLINICAL TRIAL: NCT04801823
Title: Can Early Introduction of Tree Nuts Prevent Tree Nut Allergy in Infants At High Risk of Tree Nut Allergy: the TreEat Study: a Randomised, Open-label Controlled Trial
Brief Title: The TreEat Study- Can Early Introduction of Tree Nuts Prevent Tree Nut Allergy in Infants with Peanut Allergy
Acronym: TreEat
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 70489
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Food Allergy in Infants; Nut Allergy
Keywords: food allergy; nut allergy
MeSH Terms: conditions — Nut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home Introduction of Individual tree nuts (Active Comparator): Current standard of care which is to advise families of infants diagnosed with peanut allergy to introduce tree nuts individually via a standardized, graded and cautious home introduction protocol. Day 1: smear of nut paste to the inside of lip; Day 2: 1/8 teaspoon; Day 3: 1/4 teaspoon; Day 4: 1/2 teaspoon; Day 5: 1 teaspoon. Repeat process with each individual tree nut.
  Interventions: Other: Home introduction
- In hospital multi-tree nut (almond, cashew hazelnut and walnut) oral food challenge (OFC) (Experimental): Infant will be booked for a 4-nut butter (Almond, Hazelnut, Walnut, and Cashew) graded and supervised OFC in the allergy clinical trials unit at the Murdoch Children's Research Institute. The nut butter contains a 1g dose of each nut protein in a total weight of 20g. Doses will be administered every 15minutes (1. Smear to inside of lip, 2.1/8 teaspoon, 3.1/4 teaspoon, 4.1/2 teaspoon, 5.1 teaspoon, 6.remainder of 20g nut butter paste) If challenge negative, infants continue home introduction of tree nuts as per written instructions provided. If challenge positive, infants will have additional SPT (for full tree nut panel) and single tree nut OFC as per protocol to determine tolerance/allergic status (and +/- home introduction recommendation) for each tree nut.
  Interventions: Other: Multi Nut oral food challenge

INTERVENTIONS:
Other: Home introduction — Cautious, graded introduction of individual tree nuts
  Arms: Home Introduction of Individual tree nuts
Other: Multi Nut oral food challenge — In hospital multi nut oral food challenge (almond, cashew, hazelnut, walnut)
  Arms: In hospital multi-tree nut (almond, cashew hazelnut and walnut) oral food challenge (OFC)

SUMMARY:
Early and regular ingestion of the common allergens, peanut and egg has been shown to be an effective allergy prevention strategy. It is not clear whether this is also true of tree nut allergy. Current practice in many Australian allergy clinics for children with peanut allergy (high risk of tree nut allergy), is to advise families to introduce each individual tree nut into their child's diet via a cautious home introduction protocol without prior allergy testing (screening). The safety and effectiveness of an early and regular ingestion strategy for the prevention of tree nut allergy has not been formally evaluated and it is known that around a third of children with peanut allergy develop one or more other nut allergies. This trial is a 2-armed, open-label, randomized, controlled trial (RCT) to assess the safety and efficacy of a supervised hospital based multi-tree nut (almond, cashew, hazelnut and walnut) oral food challenge (OFC) + then home introduction of the remaining tree nuts versus standard care (home introduction of all 8 tree nuts) in infants with peanut allergy to reduce the risk of developing tree nut allergy.

ELIGIBILITY:
Inclusion Criteria:

Infants aged greater than 4 months and less than 11 months of age diagnosed with IgE-mediated peanut allergy in conjunction with a positive SPT (≥3mm) or sIgE (specific immunoglobulin E) (>0.35 kU/L)

Exclusion Criteria:

* Any history of severe food induced anaphylaxis. Defined as reaction requiring 2 doses of intramuscular (IM) adrenaline.
* Pre-existing tree nut allergy (parent-reported).
* Any tree nut already tolerated (ingestion on >3 occasions without reaction of around 1 teaspoon)
* SPT or sIgE performed to any tree nuts
* Not commenced or unable to eat solid food
* Prescribed beta-blocker medication

Ages: 4 Months to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Difference between the two treatment arms in the proportion of participants with clinical confirmed tree nut allergy at 18 months of age | 18 months of age
  Tree nut allergy outcomes at 18 months will be defined as:
  1. Allergic - has evidence of tree nut sensitization (SPT>=3mm) and has had a reaction consistent with IgE (immunoglobulin E) mediated food allergy OR positive formal OFC
  2. Tree nut tolerant- successfully tolerated the tree nut at home on more than 3 occasions of at least 1 teaspoon of nut per occasion OR has had a negative formal OFC.
  3. Inconclusive -has an unknown outcome as ingestion has not occurred and participant declines OFC.

SECONDARY OUTCOMES:
Difference between the two treatment arms in the proportion of participants with ongoing peanut allergy at 18 months of age | 18 months of age
  Peanut allergy will be defined as peanut sensitization (SPT >=3mm) AND has had a reaction consistent with IgE mediated food allergy since randomization OR positive formal OFC
Difference between the two treatment arms in the proportion and severity of reported adverse events (AE) related to tree nut ingestion. | 18 months of age
  Number and severity of adverse events (AE) as assessed by standardised predetermined criteria, related to tree nut ingestion from randomization to 18 months of age collected via parent questionnaire and medical history.
Difference between the two treatment arms in the proportion and severity of solicited AEs related to tree nut ingestion. | 18 months of age
  Number and severity of solicited AEs as assessed by standardized predetermined criteria, related to tree nut ingestion from randomization to 18 months of age collected via parent questionnaire and medical history.
Difference between the 2 treatment arms in the number of tree nuts ingested. | 18 months of age
  Parent reported tree nut ingestion history based on questionnaire at baseline and 18 months of age. 0-8 tree nuts and the higher the number of tree nuts the better.
Difference between the 2 treatment arms in the frequency of tree nuts ingested. | 18 months of age
  Parent reported tree nut ingestion history based on questionnaire at baseline and 18 months of age. Range will be never to daily with higher frequency better.
Difference between the two treatment arms in mean change from baseline of Quality of Life Scores using the Food Allergy Quality of Life Questionnaire (FAQLQ-PF)- Parent Form at 18 months of age. | Baseline and 18 months of age
  The Food Allergy Quality of Life Questionnaires (FAQLQ) are disease-specific health-related quality of life (HRQL) questionnaires for patients with food allergy. FAQLQ-PF (Parent Form), completed by parents of children aged 0-12 years consists of 30 items over 3 domains (emotional impact, food anxiety, social and dietary restrictions). Total and domain scores are calculated by dividing the sum of completed items by the number of completed items. Questions are based on a 6 point Likert scale with higher scores indicating greater impact on quality of life
Difference between the two treatment arms in the mean change from baseline in State/Trait anxiety scores using the State/Trait Anxiety Inventory | Baseline and 18 months of age
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. The total score ranges from 0-63 with higher scores positively correlated with higher levels of anxiety.
Difference in the number of allergy-related healthcare visits from randomization to 18 months of age between the treatment arms | 18 months of age
  Captured per number of hospitalizations, Emergency room (ER) visits, physician office visits, and medications / number of prescriptions from randomization to 18 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Perrett, MD. PhD, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Murdoch Children's Research Institute (MCRI), Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the TreEat trial will be available six months after publication of the primary outcome. The study protocol may be obtained from the Murdoch Children's Research Institute. Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the TreEat trial investigators must see and approve the analysis plan describing how the data will be analyzed, there must be an agreement around appropriate acknowledgment and any additional costs involved must be covered. Should the study investigators be unavailable, this role is delegated to the Murdoch Children's Research Institute. Data will only be shared with a recognized research institute which has approved the proposed analysis plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication of primary outcome
Access Criteria: Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the TreEat trial investigators must see and approve the analysis plan describing how the data will be analyzed, there must be an agreement around appropriate acknowledgment and any additional costs involved must be covered.

REFERENCES:
- [Background] Ball H, Luyt D, Bravin K, Kirk K. Single nut or total nut avoidance in nut allergic children: outcome of nut challenges to guide exclusion diets. Pediatr Allergy Immunol. 2011 Dec;22(8):808-12. doi: 10.1111/j.1399-3038.2011.01191.x. Epub 2011 Sep 19. PMID 21929602
- [Background] Cifuentes L, Vosseler S, Blank S, Seismann H, Pennino D, Darsow U, Bredehorst R, Ring J, Mempel M, Spillner E, Ollert MW. Identification of Hymenoptera venom-allergic patients with negative specific IgE to venom extract by using recombinant allergens. J Allergy Clin Immunol. 2014 Mar;133(3):909-10. doi: 10.1016/j.jaci.2013.09.047. Epub 2013 Nov 28. No abstract available. PMID 24290287
- [Background] Dang TD, Mills CE, Allen KJ. Determination of the clinical egg allergy phenotypes using component-resolved diagnostics. Pediatr Allergy Immunol. 2014 Nov;25(7):639-43. doi: 10.1111/pai.12301. Epub 2014 Nov 25. PMID 25376255
- [Background] Dang TD, Tang M, Choo S, Licciardi PV, Koplin JJ, Martin PE, Tan T, Gurrin LC, Ponsonby AL, Tey D, Robinson M, Dharmage SC, Allen KJ; HealthNuts study. Increasing the accuracy of peanut allergy diagnosis by using Ara h 2. J Allergy Clin Immunol. 2012 Apr;129(4):1056-63. doi: 10.1016/j.jaci.2012.01.056. Epub 2012 Mar 3. PMID 22385632
- [Background] Ierodiakonou D, Garcia-Larsen V, Logan A, Groome A, Cunha S, Chivinge J, Robinson Z, Geoghegan N, Jarrold K, Reeves T, Tagiyeva-Milne N, Nurmatov U, Trivella M, Leonardi-Bee J, Boyle RJ. Timing of Allergenic Food Introduction to the Infant Diet and Risk of Allergic or Autoimmune Disease: A Systematic Review and Meta-analysis. JAMA. 2016 Sep 20;316(11):1181-1192. doi: 10.1001/jama.2016.12623. PMID 27654604
- [Background] Lange L, Lasota L, Finger A, Vlajnic D, Busing S, Meister J, Broekaert I, Pfannenstiel C, Friedrichs F, Price M, Trendelenburg V, Niggemann B, Beyer K. Ana o 3-specific IgE is a good predictor for clinically relevant cashew allergy in children. Allergy. 2017 Apr;72(4):598-603. doi: 10.1111/all.13050. Epub 2016 Nov 17. PMID 27644013
- [Background] McWilliam V, Peters R, Tang MLK, Dharmage S, Ponsonby AL, Gurrin L, Perrett K, Koplin J, Allen KJ; HealthNuts investigators. Patterns of tree nut sensitization and allergy in the first 6 years of life in a population-based cohort. J Allergy Clin Immunol. 2019 Feb;143(2):644-650.e5. doi: 10.1016/j.jaci.2018.07.038. Epub 2018 Aug 30. PMID 30171872
- [Background] Mullins RJ, Wainstein BK, Barnes EH, Liew WK, Campbell DE. Increases in anaphylaxis fatalities in Australia from 1997 to 2013. Clin Exp Allergy. 2016 Aug;46(8):1099-110. doi: 10.1111/cea.12748. Epub 2016 May 31. PMID 27144664
- [Background] Pablos I, Wildner S, Asam C, Wallner M, Gadermaier G. Pollen Allergens for Molecular Diagnosis. Curr Allergy Asthma Rep. 2016 Apr;16(4):31. doi: 10.1007/s11882-016-0603-z. PMID 27002515
- [Background] Peters RL, Barret DY, Soriano VX, McWilliam V, Lowe AJ, Ponsonby AL, Tang MLK, Dharmage SC, Gurrin LC, Koplin JJ, Perrett KP. No cashew allergy in infants introduced to cashew by age 1 year. J Allergy Clin Immunol. 2021 Jan;147(1):383-384. doi: 10.1016/j.jaci.2020.07.003. Epub 2020 Jul 18. No abstract available. PMID 32693093
- [Background] Sampson HA, Gerth van Wijk R, Bindslev-Jensen C, Sicherer S, Teuber SS, Burks AW, Dubois AE, Beyer K, Eigenmann PA, Spergel JM, Werfel T, Chinchilli VM. Standardizing double-blind, placebo-controlled oral food challenges: American Academy of Allergy, Asthma & Immunology-European Academy of Allergy and Clinical Immunology PRACTALL consensus report. J Allergy Clin Immunol. 2012 Dec;130(6):1260-74. doi: 10.1016/j.jaci.2012.10.017. No abstract available. PMID 23195525
- [Background] Savvatianos S, Konstantinopoulos AP, Borga A, Stavroulakis G, Lidholm J, Borres MP, Manousakis E, Papadopoulos NG. Sensitization to cashew nut 2S albumin, Ana o 3, is highly predictive of cashew and pistachio allergy in Greek children. J Allergy Clin Immunol. 2015 Jul;136(1):192-4. doi: 10.1016/j.jaci.2015.03.037. Epub 2015 May 8. No abstract available. PMID 25959668
- [Background] Soriano VX, Peters RL, Ponsonby AL, Dharmage SC, Perrett KP, Field MJ, Knox A, Tey D, Odoi S, Gell G, Camesella Perez B, Allen KJ, Gurrin LC, Koplin JJ. Earlier ingestion of peanut after changes to infant feeding guidelines: The EarlyNuts study. J Allergy Clin Immunol. 2019 Nov;144(5):1327-1335.e5. doi: 10.1016/j.jaci.2019.07.032. Epub 2019 Aug 8. PMID 31401287
- [Background] Thalayasingam M, Noble V, Franzmann A, O'Sullivan M. Outcome of mixed nut biscuit challenges in low-risk patients who are on tree nut exclusion diet. Pediatr Allergy Immunol. 2015 Nov;26(7):682-4. doi: 10.1111/pai.12437. Epub 2015 Sep 11. No abstract available. PMID 26126774
- [Background] Togias A, Cooper SF, Acebal ML, Assa'ad A, Baker JR Jr, Beck LA, Block J, Byrd-Bredbenner C, Chan ES, Eichenfield LF, Fleischer DM, Fuchs GJ 3rd, Furuta GT, Greenhawt MJ, Gupta RS, Habich M, Jones SM, Keaton K, Muraro A, Plaut M, Rosenwasser LJ, Rotrosen D, Sampson HA, Schneider LC, Sicherer SH, Sidbury R, Spergel J, Stukus DR, Venter C, Boyce JA. Addendum guidelines for the prevention of peanut allergy in the United States: Report of the National Institute of Allergy and Infectious Diseases-sponsored expert panel. J Allergy Clin Immunol. 2017 Jan;139(1):29-44. doi: 10.1016/j.jaci.2016.10.010. PMID 28065278
- [Background] van der Valk JPM, Bouche RE, Gerth van Wijk R, de Groot H, Wichers HJ, Dubois AEJ, de Jong NW. Low percentage of clinically relevant pistachio nut and mango co-sensitisation in cashew nut sensitised children. Clin Transl Allergy. 2017 Mar 20;7:8. doi: 10.1186/s13601-017-0145-z. eCollection 2017. PMID 28321292
- [Background] Van Erp FC, Knulst AC, Kok IL, van Velzen MF, van der Ent CK, Meijer Y. Usefulness of open mixed nut challenges to exclude tree nut allergy in children. Clin Transl Allergy. 2015 May 16;5:19. doi: 10.1186/s13601-015-0062-y. eCollection 2015. PMID 26034579
- [Background] Zahradnik E, Raulf M. Respiratory Allergens from Furred Mammals: Environmental and Occupational Exposure. Vet Sci. 2017 Aug 4;4(3):38. doi: 10.3390/vetsci4030038. PMID 29056697
- [Derived] McWilliam VL, Koplin JJ, Allen K, Robinson M, Smart J, Loke P, Peters RL, Dang T, Lee KJ, Dalziel K, Tey D, Taranto M, Perrett KP. TreEAT trial: Protocol for a randomized controlled trial investigating the efficacy and safety of early introduction of tree nuts for the prevention of tree nut allergy in infants with peanut allergy. Pediatr Allergy Immunol. 2023 Mar;34(3):e13930. doi: 10.1111/pai.13930. PMID 36974653